CLINICAL TRIAL: NCT03838172
Title: The Effects of Burn Injury on Parents
Brief Title: Investigation of the Impact of Burn Injury on Parents
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozden Ozkal, Principal Investigator, Hacettepe University
Other Study IDs: GO 19/28
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Burns; Parents
Keywords: Burn Injury; quality of life; scar
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: Parents who have a burned child
  Interventions: Other: Family impact scale

INTERVENTIONS:
Other: Family impact scale — The family Impact Scale (FIS) will be completed by the parents

SUMMARY:
Burn injuries are related to longer hospital stay. Patients who have a burned child are affected prolonged hospitalization. Social life and quality of life are affected by burn injuries. Therefore, the aim of this study is to investigate the effects of burn injury on parents.

DETAILED DESCRIPTION:
Pediatric burn injuries is commonly seen. Burn injuries are extended from minor injuries to severe injuries. The severity of burn injury may affect burn related complications such as scar tissue and duration of hospitalization. This process extremely affect parents. Although parents are part of this prolonged treatments process, there is no study that evaluated of the impact of burn injury on parents. Therefore, the aim of this study is to investigate the effects of burn injury on parents.

ELIGIBILITY:
Inclusion Criteria:

* Parents who have a burned child
* Parents who have a volunteer

Exclusion Criteria:

* Parents who have no confirm to participate this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents who have a burned child
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Family of Impact scale | 15 minutes
  questionnaire is a self-report instrument designed to measure the effects of childhood diseased on parents. A low score indicates a higher impact of the disease on the parents.

SECONDARY OUTCOMES:
Nottingham Health Profile | 15 minutes
  Nottingham Health Profile is a widely used measure of perceived health status. The higher score is indicated the lower quality of life.
The hospital anxiety and depression scale | 15 minutes
  It is a self-reported questionnaire that measures level of anxiety and depression. the higher score is indicated the higher anxiety level.
The Spielberger State-Trait Anxiety Inventory | 15 minutes
  It is used to determine anxiety level of parents. Higher scores are an indication of greater anxiety.
Patient and Observer Scar Assessment Scale | 15 minutes
  The Patient and Observer Scar Assessment Scale consists of two scales, the patient scale, which contains six items, and the observer scale, which contains five items. The higher score indicates the greater scar tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Ozden Ozkal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No